CLINICAL TRIAL: NCT05771792
Title: Comparison of Eccentric Training on Injury Prevention and Hamstring Strength in Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01404 Shivam Sachdev
Record Dates: First submitted 2023-01-13; First posted 2023-03-16 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Sport Injury; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eccentric exercise group (Experimental): SPECIFIC MODIFIED EXERCISE PROGRAM GROUP The modified exercise group will perform 6 exercises
  Interventions: Other: ECCENTRIC EXERCISE
- control group (Active Comparator): CONVENTIONAL EXERCISES PROGRAM GROUP The conventional exercises program will perform conventional exercises.
  Interventions: Other: CONVENTIONAL EXERCISES PROGRAM

INTERVENTIONS:
Other: ECCENTRIC EXERCISE — Eccentric Exercise training group will perform 8 weeks of protocol with a total 24 sessions for 45 minutes (3 session per week). During each 45 minutes training session, subjects will complete the warmup for 10 minutes, Eccentric Exercise training for 25 minutes and cool down 10minutes. All players will perform each repetition in a slow, controlled manner, 10 repetition and 3 sets in first 4 week and 15 repetition and 3 sets in last 4 weeks of all exercises for 45 minutes. Eccentric exercise training protocol is as follow: Prone Hamstring Curl, Seated TheraBand Hamstring Curl, Exercise Ball (or glider) Bridge with Curl, Stiff-Legged Deadlift, Single Leg Deadlift, Nordic Hamstring Curl.
  Arms: eccentric exercise group
Other: CONVENTIONAL EXERCISES PROGRAM — The participant of the Control Group will perform 8 weeks of protocol with a total 24 sessions for 45 minutes (3 session per week). During each 45 minutes training session, subjects will complete the warmup for 10 minutes, conventional training for 25 minutes and cool down 10minutes. All players will perform each repetition in a slow, controlled manner, 10 repetition and 3 sets in first 4 week and 15 repetition and 3 sets in last 4 weeks of all exercises for 45 minutes. The exercise will be as follow: Side Lunges, Split Squats, Calf Raises.
  Arms: control group

SUMMARY:
To determine the effect of the eccentric exercise training on injury prevention and hamstring strength in football players.

DETAILED DESCRIPTION:
Hamstrings injuries are common among footballers with a higher prevalence rate in male footballers. Despite the relatively high incidence of hamstring injuries in sports, no clear prevention methods have been identified. Most hamstring muscle injuries occur during an eccentric phase of any activity. Eccentric hamstring training has been used for injury prevention in recent years. The two distinguishing characteristics of eccentric muscle contractions have been well understood: 1) great force output; and 2) low energy cost to produce the force. Due to these distinguishing characteristics, eccentric exercise is widely used in injury prevention programs.

The aim of this study is to determine the effectiveness of eccentric training as compared to conventional training in hamstring muscle injury prevention and strengthing in football players.

ELIGIBILITY:
Inclusion Criteria:

* Football players with age 18 to 40
* Male
* Players playing football for > 1 year

Exclusion Criteria:

* Having history of injury and surgery in past
* Those players having any kind of musculoskeletal, neurological, cardiovascular, or degenerative problems
* Those players who have any medical conditions

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Hamstring Strength | 8 weeks
  Vertical jumps: The person puts chalk on their finger tips to mark the wall at the height of their jump. The person then stands away from the wall, and jumps vertically as high as possible using both arms and legs to assist in projecting the body upwards. Attempt to touch the wall at the highest point of the jump.
Anaerobic Capacity | 8 weeks
  SPRINT FATIGUE TEST: A repeat sprint test of anaerobic capacity consisting of ten 30-second sprints. This is an anaerobic capacity test, which measures the ability to recover between sprints while maintaining the same level of strength.
Agility | 8 weeks
  5-0-5 AGILITY TEST: The ability to turn 180 degrees is measured by the 505 Agility test. The test can also be modified for sport-specific testing by having the subject dribble a soccer ball, a hockey puck, or a basketball through the course.

SECONDARY OUTCOMES:
Injury Prevention ( FASH ) | 8 weeks
  FASH (Functional assessment scale for acute hamstring injuries) questionnaire is a self-administered questionnaire used for acute hamstring injuries assessment. It is a valid and reliable instrument for assessing and determining the severity of hamstring injuries in an athlete population. It is a 10-item questionnaire that look the ability of a patient to perform certain lower extremity activities. This is a self-report questionnaire that patient can rate difficulty and interference with daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Saad Rauf, Ph.D*, Principal Investigator — Riphah International University
Locations (1):
- Etihad Football Club, Quetta, Balochistan, Pakistan

IPD SHARING:
Plan to Share IPD: No